CLINICAL TRIAL: NCT04735380
Title: Agreements Between Transcutaneous and Arterial Monitoring of Oxygen and Carbon Dioxide After Non-cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Eske Kvanner Aasvang, Clinical professor, Rigshospitalet, Denmark
Other Study IDs: P-2020-1159
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Post Anesthesia Care Optimaization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: TCM-5 Flex monitor connected to a Sensor 84 (Radiometer Medical Aps, Brønshøj, Denmark) — Patients undergo 2-3 hrs of observation while wearing the device.

SUMMARY:
The primary aim of the study is to describe the association between changes in TcO2 and TcCO2 and interventions such as blood transfusion, fluid therapy, respiratory support, use of vasopressors, analgesics, and adverse events during PACU admission. The secondary aim is to describe the agreement between TcPO2 and TcPCO2 and PaO2 and PaCO2 in patients after non-cardiac surgery.

DETAILED DESCRIPTION:
Study method The data collection will start 1st of February 2021 and will be finished by 30th of April 2021. Patients will be set up with TCM equipment and an Empatica at the PACU. They will be observed for 2 hours. If an intervention is started before 2 hours and not completed, recordings will continue until 5 minutes after the intervention is completed for a maximum of 1 hour (3 hours maximal observation). The sensor will be placed on the patient's antebrachium. Patients will be set up with TCM equipment as soon as possible after arrival at PACU. Every clinical procedure entailing changes in circulatory and/or respiratory support or medication (appendix 1) will be observed and noted in a timetable (ap-pendix 2). Perfusion index (PI) and a full DASAIM score (Danish Association of Anesthesiology and Intensive Care Medicine) will be noted every 15 minutes. Every ABG analysis of PaO2, PaCO2 and lactate conducted during the observational period will be noted.

Age, sex, BMI (Body Mass Index), ASA-score (American Society of Anesthesiologists physical sta-tus classification), comorbidity (Charlson Comorbidity Index - CCI), baseline laboratory data (hemo-globin and creatinine) and name of surgical procedure will be obtained for each patient. REDCap (Research Electronic Data Capture) will be used as a data management system for the project. The study is a part of the Wireless Assessment of Respiratory and circulatory Distress (WARD) project.

Study materials All patients will be monitored with a TCM-5 Flex monitor connected to a Sensor 84 (Radiometer Medical Aps, Brønshøj, Denmark). The sensor consists of a Stow-Severinghaus-type TcPCO2 electrode combined with a Clark-type TcPO2 electrode, with values per second for TcPO2, TcPCO2 in kPa and heat effect measured in units of mW. The sensor temperature will automatically be heated to 43.5℃ and calibrated. The sensor membrane will be changed every 28th day. There will be a 20-minute stabilization period from patient setup to valid data capturing. The use of sensors and monitors will be according to the manufacturer's instructions.

As a supplement, patients will be wearing an Empatica, as a measurement for the activity of the autonomic nervous system. The Empatica tracks activity, heartrate, blood volume pulse, skin temper-ature and skin conductance. The Empatica E4 consist of a PPG sensor and an EDA sensor. Data from the E4 will be processed in further studies and is not a part of the statistical analysis in this protocol.

Statistics The primary analysis is changes in TCM readings, and the association between clinical procedures, tested using paired statistics comparing both average (mean) TcPO2 and TcPCO2 during 5 minutes before an intervention versus 5 minutes after an intervention. Depending on the data distribution, either t-test or Wilcoxon test will be used.

Secondary analysis includes:

* Changes in TCM and association with specific intervention including grouping into circulatory and respiratory groups.
* Agreement between TcPO2 and PaO2, TcPCO2 and PaCO2. Agreement between the two tech-niques will be assessed using Bland-Altmann analysis including description of mean differ-ence and limits of agreement(17). In case of left-skewed data, log transformation will be ap-plied. A four-quadrant plot will be constructed to assess trending ability and a concordance rate will be calculated.

Tertiary analysis includes:

* An ANCOVA (analyses of co-variance) of the primary and secondary outcomes, with the following predefined variables: age, sex, BMI, ASA-score, and comorbidity, baseline labora-tory data (hemoglobin and creatinine).
* Agreement between perfusion-index and TCM. Agreement between the two techniques will be assessed using Bland-Altmann analysis including description of mean difference and limits of agreement. In case of left-skewed data, log transformation will be applied. A four-quadrant plot will be constructed to assess trending ability and a concordance rate will be calculated.

All results will be stated with their 95% confidence interval (CI). The significance level will be 5%, meaning p-values under 0.05 will be acknowledged as statistically significant. All analyses will be performed using Python 3.7 and the software program PyCharm.

ELIGIBILITY:
Inclusion Criteria:

* A scheduled stay at PACU for at least 3 postoperatively.

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be patients undergoing major abdominal, urological, vascular, or orthope-dic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
TCM changes | 31-08-21
  The primary outcome is changes in TCM recordings before and after clinical interventions and/or acute severe adverse events.

SECONDARY OUTCOMES:
ABG and TCM | 31-08-21
  The secondary outcome is changes in arterial blood gasses before and after clinical interventions and/or acute severe adverse events if recorded in the PACU.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thy SA, Johansen AO, Thy A, Sorensen HH, Molgaard J, Foss NB, Toft P, Meyhoff CS, Aasvang EK. Associations between clinical interventions and transcutaneous blood gas values in postoperative patients. J Clin Monit Comput. 2023 Oct;37(5):1255-1264. doi: 10.1007/s10877-023-00982-x. Epub 2023 Feb 18. PMID 36808596